CLINICAL TRIAL: NCT03062007
Title: Open-label Study of Safety, Tolerability and Pharmacokinetics of Multiple Doses of BI-CON-02 in Patients With HER2-positive Metastatic Breast Cancer, Previously Treated With Trastuzumab
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Biointegrator LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-BICON02-01
Record Dates: First submitted 2017-02-08; First posted 2017-02-23 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI-CON-02 (Experimental): The start dose of BI-CON-02 will be 0,3 mg/kg and it will be possible to increase gradually BI-CON-02 doses up to 0,6 mg/kg; 1,2 mg/kg; 2,4 mg/kg; 3,6 mg/kg and 4,8 mg/kg for subsequent dose cohorts. A possibility to include a new dose cohort in the study will be considered by the Data and Safety Monitoring Committee, basing on the data of BI-CON-02 safety and tolerability, received at the Visit (Week 3, Day1) in the previous dose cohort (3 weeks after - 21st day of therapy).
  Interventions: Drug: BI-CON-02

INTERVENTIONS:
Drug: BI-CON-02 — BI-CON-02 prescribed as intravenous infusion once per 3 weeks. Investigational product therapy during 1 year (up to 18 cycles, duration of 21 days each).

SUMMARY:
This study will evaluate the safety and tolerability of BI-CON-02 in patients with HER2-positive metastatic breast cancer, previously treated with trastuzumab The clinical trial protocol for BI-CON-02 prescribes a start dose of 0,3 mg/kg. After the Data and Safety Monitoring Committee evaluates the data of tolerability and safety of BI-CON-02, received during 3 weeks of investigational product therapy (Week 3, Day 1) and approves, extra doses can be used.

Once the safety of investigational product is confirmed, the dose will be increased in the subsequent cohorts. Planned doses - 0,3 mg/kg; 0,6 mg/kg; 1,2 mg/kg; 2,4 mg/kg; 3,6 mg/kg and 4,8 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

To participate in the clinical study, patients must comply to the following criteria:

1. Signed patient's information sheet and informed consent form to participate in the study
2. Females aged ≥ 18 years
3. Histologically confirmed diagnosis of locally advanced or metastatic breast cancer.
4. HER2-positive tumor status by results of immunohistochemistry (IHC3+) or hybridization in-situ (ISH), received at the local laboratory, experienced/certified to determine HER2 expression by means of accurate and validated methods.
5. Disease progression during or after trastuzumab-based chemotherapy.
6. Previous chemotherapy on metastatic breast cancer.
7. Requirements for laboratory parameters determined below:

   Hematology: Absolute neutrophil count:

   Platelets:

   Hemoglobin: ≥ 1500/mm3 (1.5 x 109 cells/L)
   * 100 000/mm3 (100 x 109 cells/L)
   * 9.0 g/dl

   Liver function: Total bilirubin:

   Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkalinephosphatase ≤ 1.5 x ULN

   ≤ 2.5 x ULN or ≤ 5.0 х ULN in case of liver and/or bones metastasis Renal function: Serum creatinine or GFR (according to Cocroft-Golt formula): ≤ 1.5 mg/dl > 60 ml/min
8. Patients must have an ECOG status of 0, 1 or 2
9. Women of childbearing potential (not sterile or in menopause less than 2 years) must be practicing an effective method of birth control during the whole period of the study and 6 months after the last administration of the investigational product. Effective methods of birth control include usage of a condom or diaphragm (barrier method) with spermicide.

Exclusion Criteria:

The patient will be considered ineligible for the study in case she has any criteria listed here below:

1. Clinically significant cardiovascular diseases:

   * Myocardial infarction within 6 months before screening
   * Unstable angina within 3 months before screening
   * Congestive heart failure Class III or IV according to the New York Heart Association (NYHA) criteria
   * Clinically significant ventricular arrhythmia, that have to be treated, including ventricular tachycardia, ventricular fibrillation, history of cardiac arrest
   * QTc interval > 460 ms (ECG) (calculated according to Fredericia formula), or a diagnosis of long QTc syndrome
   * Ejection fraction of left ventricle ≤ 50% (EchoCG)
   * Hypotension (systolic arterial blood pressure < 86 mm of mercury) or bradycardia with a heart rate of < 50 beats per min., except when caused by medications (e.g. beta-blockers)
   * Uncontrolled arterial hypertension (systolic arterial blood pressure > 170 mm of mercury or diastolic arterial blood pressure > 105 mm of mercury)
   * Troponins I ≥ 0.2 ng/ml
2. Patients with known cerebral metastases or clinical signs of cerebral metastases.
3. Patients with severe dyspnea at rest, or those who need additional oxygen therapy in everyday life.
4. History of hypersensitivity to trastuzumab ≥ 3 severity level
5. History of any toxicity related to trastuzumab administration that resulted in the termination of trastuzumab therapy.
6. Peripheral neuropathy ≥ II severity level
7. Bisphosphonate therapy for symptomatic hypercalcemia.
8. Any chemotherapy, hormonotherapy, radiotherapy, immunotherapy or biological products therapy used for breast cancer treatment within 4 weeks before the first administration of the investigational product.
9. Previous indication of doxorubicin in maximum cumulated dose > 360 mg/kg2, or its equivalent.
10. Participation in other clinical studies or administration of other investigational products within 4 weeks before the first administration of the investigational product, or presence of on-going toxicities ≥ II grade according to CTCAE, related to any prior antitumour therapy (excluding alopecia).
11. History of other malignancies with the exception of cervical carcinoma in situ or skin basal-cell carcinoma, that had undergone surgical removal and treatment within ≥ 5 years before the first administration of the investigational product.
12. Presence of antibodies to human immunodeficiency virus (HIV), or hepatitis С virus (HCV), presence of HBsAg
13. Active infection within 4 weeks before the first administration of the investigational product.
14. Uncontrolled concomitant diseases and conditions, including mental or social, which, in the Investigator's opinion, may prevent the patient from participation in the study.
15. Drug or alcohol abuse on the moment of screening or in the past, which, in the Investigator's opinion, makes the patient unsuitable for participation in the study.
16. Pregnant or lactating women, or women who plan to get pregnant during the clinical study
17. Inability to read or write, unwillingness to understand and comply with the procedures of the study protocol, as well as any other concomitant medical or serious mental conditions, that make the patient unsuitable for participation in the clinical study, limit the validity of informed consent receipt or may affect the patient's ability to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) Safety and tolerability of multiple doses of Safety and tolerability of multiple doses of BI-CON-02 | Up to Week 55
  The number of patients with treatment-related AEs assessed by CTCAE, abnormal laboratory values and instrumental tests (ECG).
Maximum tolerated dose (MTD) or recommended dose (RD) of BI-CON-02 | At Week 3 Day 1
  MTD is defined as maximum dose at which DLT occurs in more than 1 patient of 6

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Up to 55 weeks
  PK analysis of multiple doses of BI-CON-02
Immunogenetics of BI-CON-02 | Up to Week 55
  Assessment of Antibodies to BI-CON-02 in blood samples
Peak Plasma Concentration (Cmax) | Up to 55 weeks
  PK analysis of multiple doses of BI-CON-02
Elimination half-life (T1/2) | Up to 55 weeks
  PK analysis of multiple doses of BI-CON-02
Volume of distribution at steady state (Vss) | Up to 55 weeks
  PK analysis of multiple doses of BI-CON-02
Clearance (CL) | Up to 55 weeks
  PK analysis of multiple doses of BI-CON-02

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - 3. State Medical Preventive Institution "Kirov Region Clinical Oncological Dispensary", Kirov
  - 5. State Budgetary Public Healthcare Institution "Leningrad Region Oncological Dispensary", department of surgery, Leningrad Region Settlement Kuz'molovsky
  - 1. Federal State Budgetary Institution "Russian Oncological Scientific Center n.a. N.N.Blokhin" of the Russian Academy of Medical Sciences., Moscow
  - 2. Moscow State Public Healthcare Institution "Moscow City Oncological Hospital #62 of the Moscow Public Healthcare Department", Moscow Region, Krasnogorsk District, Settlement Istra
  - 6. State Budgetary Public Healthcare Institution of the Nizhni Novgorod Region "Nizhni Novgorod Region Oncological Dispensary", Nizhny Novgorod
  - 4. State Budgetary Educational Institution of Higher Professional Education "Saint-Petersburg State Medical University n.a. academician I.P.Pavlov of the Federal Agency for Public Healthcare and Social Development", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No